CLINICAL TRIAL: NCT06178016
Title: The Effect of Bystander Intervention Program on Bystander Efficacy, Behavior and Intent to Help for Dating Violence in Nursing Students
Brief Title: Efficacy of Bystander Intervention Program in Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Seda Er, Research Assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IU-Cerrahpaşa (IUC)
Record Dates: First submitted 2023-12-02; First posted 2023-12-20 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Bystander Effect; Dating Violence; Nursing Students; Intimate Partner Violence
Keywords: Bystander Intervention; Dating Violence; Nursing Students

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Participants in this group will have the Bystander Intervention Program for Dating Violence. The aim of this program, which will be prepared taking into account the needs of the country and institutions, is to provide knowledge and skills to safely intervene in dating violence. The program will be implemented at a convenient time for the experimental group of students within the 2023-2024 Spring semester academic calendar, taking into account the 1st-grade course schedule of Istanbul University-Cerrahpaşa Florence Nightingale Faculty of Nursing.
  Interventions: Other: Bystander Intervention Program for Dating Violence
- Control Group (No Intervention): The control group will not participate in the Bystander Intervention Program for Dating Violence, an interview consisting of one session is planned considering for the placebo effect. The control group students will be given a single 60-minute information session on dating violence and the students will be expected to fill out the scales to be filled out within the scope of the research at the pre-test and post-test times. At the end of the study, the Bystander Intervention Program for Dating Violence will be carried out with the voluntary participants in the control group, taking into account the ethics.

INTERVENTIONS:
Other: Bystander Intervention Program for Dating Violence — The Bystander Intervention Program for Dating Violence includes the following topics: Dating violence and its types (Session 1), risk factors and consequences of dating violence (Session 2), bystander intervention in dating violence and barriers to intervention (Session 3), bystander intervention strategies for dating violence (Session 4), self-care for bystanders witnessing dating violence (Session 5).
  Each session is planned to last 60-90 minutes. Materials will be used in the Bystander Intervention Program for Dating Violence are PPT (PowerPoint Presentations) slides, videos, interactive scenarios, and group discussions. The Bystander Intervention Program for Dating Violence is planned to be applied face-to-face in 4 groups (12, 10, and 10 people) at scheduled times in a quiet room suitable for the group.
  Arms: Experimental Group

SUMMARY:
The research will be conducted in a randomized control group experimental research design. The study aims to evaluate the effectiveness of the bystander intervention program developed for dating violence in nursing students. The Bystander Intervention Program will be developed after a literature review on the subject and taking into account previous evidence-based research. The population of the study will consist of Istanbul University-Cerrahpaşa Florence Nightingale Faculty of Nursing, Department of Nursing, Turkish Program 1st year students (N=130). In the sample size calculation, the data reported in similar studies in the literature were used (Rothman et al. 2018). The representativeness of the study was calculated as β=80%, α=0.05 (effect size: 0.6), and a total of 80 samples were calculated as a result of power analysis, 40 intervention, and 40 control groups. Participants will be assigned to the experimental or control group by computer-based simple randomization method. Data will be collected between September, 19 2024, and December 19, 2024. Data will be collected face-to-face using the Individual Information Form, Bystander Efficacy Scale, Intention to Help Scale-Short Version, Bystander Behavior Scale (For Friends), and Program Evaluation Form. The data obtained from the research will be evaluated with the SPSS package program.

DETAILED DESCRIPTION:
Dating violence is defined as the tendency to force a person, to establish power and control over a person. Dating violence is a public health problem for all countries in the world (WHO, 2021; Kerman & Öztürk, 2022). According to the results of studies conducted with university students; more than 70% of students are exposed to dating violence (Schuster et al., 2016; Toplu-Demirtaş & Fincham, 2020). In addition, it is stated in studies that dating violence starts before the age of 25 (Peterson et al., 2018; Park & Kim, 2021). Young people exposed to violence may have difficulty seeking help, hide the violence, and feel obliged to maintain the relationship (Park & Kim, 2021). Studies have shown that college students exposed to dating violence experience many negative physical and mental problems, including physical injuries, depression, anxiety, decreased academic performance, and drug and alcohol abuse (Choi et al., 2017).

One of the ways to reduce the risk of dating violence is to focus on other bystanders. It is seen that programs developed to prevent violence are shaped around bystander intervention (Banyard et al., 2019). Bystander intervention, an evidence-based intervention to prevent dating violence, is defined as "an initiative that focuses on adolescents or young adults who have the necessary skills and self-efficacy to safely intervene when they witness dating violence and sexual violence" (Storer, 2016). Bystanders can contribute to risk reduction directly (e.g. by calling security, intervening directly) or indirectly (e.g. by challenging negative attitudes towards dating violence) when dating violence occurs (Amar et al., 2015; Banyard et al., 2019; Debnam and Mauer, 2019; Finnie et al., 2022). Recent studies have found that bystander intervention programs applied to young people produce statistically significant results in the areas of (1) knowledge about dating violence (prevalence, definitions, etc.); (2) attitudes towards dating violence (decrease in sexist attitudes, decrease in denial of violence as a problem, increase in confidence to intervene, increase in intention to intervene, increase in students' self-efficacy to take action against violence, etc.) and (3) behavioral change (decrease in violence perpetration rate, etc.) (Amar et al. 2015; Jouriles et al. 2018; Peterson et al. 2018). ) and (3) behavior change (decreased rate of violence perpetration, etc.) (Amar et al. 2015; Jouriles et al. 2018; Peterson et al. 2018).

Nurses are one of the first intervention health professionals in the care of individuals exposed to violence. Providing direct care to the individual subjected to violence and advocating for resources focused on preventing violence is one of the responsibilities and roles of nursing care. It is stated that mental health nurses can apply bystander education principles in prevention programs that aim to change community norms regarding violence (Amar et al. 2012; Kerman & Öztürk, 2022). It is stated that it is important for nursing students, who will be among the health professionals of the future, to develop knowledge, skills, and attitudes about what to do when they witness violence (Barroso-Corroto ve ark., 2022). There are different bystander intervention programs used to prevent dating violence in the literature (Debnam & Mauer, 2019). However, there is no bystander intervention program developed for dating violence for university students in Turkey. Accordingly, this study aims to evaluate the effectiveness of the bystander intervention program developed for dating violence in nursing students.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-24
* Active student enrollment in the nursing department of the faculty in the academic year 2023-2024
* Filled in forms and scales

Exclusion Criteria:

* No active student enrollment in the nursing department of the faculty in the academic year 2023-2024 (due to reasons such as freezing enrollment, transferring to another institution, etc.)
* Participation in seminars/workshops/group work/conferences/congresses/seminars/trainings etc. on prevention of dating violence and/or bystander intervention

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-06-13 (Actual)

PRIMARY OUTCOMES:
Bystander Efficacy Scale | It will be applied to both groups within one week before the program, and within 1 week after the program is completed
  The scale used to assess bystander effectiveness was developed by Banyard et al. The scale includes 18 items. The participant is expected to indicate his/her degree of confidence by writing a whole number between 0-100 to indicate how confident he/she is that he/she can perform the behaviors specified in the scale. The calculation is made by averaging all items and the scale has no cut-off point. High scores indicate a high degree of confidence. In the study conducted by Banyard et al. (2014), the Cronbach's alpha value of the scale was .93 and the mean was 72.60.
Intention to Help Scale-Short Version | It will be applied to both groups within one week before the program, and within 1 week after the program is completed
  The scale, which assesses the likelihood or willingness of participants to engage in various helping behaviors, was developed by Banyard et al. (2014). There are two separate subscales by creating separate but parallel items and it consists of 18 items in total. Participants are expected to rate their likelihood of performing the behaviors using a 5-point Likert-type scale. The scale is calculated by averaging the answers given to the items. High scores indicate that the individual is more likely to engage in helping behavior. Cronbach's alpha value for the short version of the scale was .93 (Banyard et al. 2014).
Bystander Behavior Scale (For Friends) | It will be applied to both groups 2 months after the program
  The scale used to determine the spectator behavior of the participants in the last 2 months was developed by Banyard et al. The scale has 44 items and includes only spectator behaviors towards friends. The scale consists of 4 factors. Participants are expected to mark "Yes", "No" and "Did not meet" for the fulfillment of each item. In the evaluation, each no sign is calculated as 0 points and each yes sign is calculated as 1 point. The items that individuals said they did not encounter are not included in the scoring and the calculation is made by taking the average of the answers given to the other items. Higher scores indicate the types of bystander behavior reported by more people. Cronbach's alpha value for the short version of the scale was .971 (Banyard et al. 2014).

CONTACTS AND LOCATIONS:
Overall Officials: Sevim Buzlu, PhD,RN, Study Chair — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpaşa, Istanbul, Şişli/Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD (Individual Participant Data) available. After the study is completed, the publication which includes the data results will be available.

REFERENCES:
- [Background] Rothman EF, Paruk J, Banyard V. The escalation dating abuse workshop for college students: Results of an efficacy RCT. J Am Coll Health. 2018 Aug-Sep;66(6):519-528. doi: 10.1080/07448481.2018.1431909. Epub 2018 Mar 22. PMID 29405867
- [Background] Storer HL, Casey E, Herrenkohl T. Efficacy of Bystander Programs to Prevent Dating Abuse Among Youth and Young Adults: A Review of the Literature. Trauma Violence Abuse. 2016 Jul;17(3):256-69. doi: 10.1177/1524838015584361. Epub 2015 May 6. PMID 25951840
- [Background] Debnam KJ, Mauer V. Who, When, How, and Why Bystanders Intervene in Physical and Psychological Teen Dating Violence. Trauma Violence Abuse. 2021 Jan;22(1):54-67. doi: 10.1177/1524838018806505. Epub 2019 Jan 22. PMID 30669950
- [Background] Banyard VL, Moynihan MM, Cares AC, Warner R. How do we know if it works? Measuring outcomes in bystander-focused abuse prevention on campuses. Psychology of Violence. 2014;4(1):101.
- [Background] Banyard V, Moschella E, Grych J, Jouriles E. What happened next? New measures of consequences of bystander actions to prevent interpersonal violence. Psychology of Violence. 2019; 9(6):664-674.
- [Background] Tekkas Kerman K, Ozturk FO. An examination of gender stereotypes, ambivalent sexism, and dating violence as potential predictors of nursing students' beliefs about intimate partner violence: A cross-sectional correlational study. Nurse Educ Pract. 2022 Jul;62:103346. doi: 10.1016/j.nepr.2022.103346. Epub 2022 Apr 6. PMID 35430535
- [Background] Schuster I, Krahe B, Toplu-Demirtas E. Prevalence of Sexual Aggression Victimization and Perpetration in a Sample of Female and Male College Students in Turkey. J Sex Res. 2016 Nov-Dec;53(9):1139-1152. doi: 10.1080/00224499.2016.1207057. Epub 2016 Aug 2. PMID 27485372
- [Background] Toplu-Demirtas E, Fincham FD. I Don't Have Power, and I Want More: Psychological, Physical, and Sexual Dating Violence Perpetration Among College Students. J Interpers Violence. 2022 Jul;37(13-14):NP11490-NP11519. doi: 10.1177/0886260520951319. Epub 2020 Aug 25. PMID 32840154
- [Background] Park S, Kim SH. A mixed-method pilot study to test a program for friend-supporters of victims of dating violence. J Community Psychol. 2021 Jul;49(5):1153-1168. doi: 10.1002/jcop.22568. Epub 2021 Mar 29. PMID 33778972
- [Background] Peterson K, Sharps P, Banyard V, Powers RA, Kaukinen C, Gross D, Decker MR, Baatz C, Campbell J. An Evaluation of Two Dating Violence Prevention Programs on a College Campus. J Interpers Violence. 2018 Dec;33(23):3630-3655. doi: 10.1177/0886260516636069. Epub 2016 Mar 13. PMID 26976433
- [Background] Choi EP, Wong JY, Fong DY. Mental health and health-related quality of life of Chinese college students who were the victims of dating violence. Qual Life Res. 2017 Apr;26(4):945-957. doi: 10.1007/s11136-016-1413-4. Epub 2016 Sep 22. PMID 27660071
- [Background] Finnie RKC, Okasako-Schmucker DL, Buchanan L, Carty D, Wethington H, Mercer SL, Basile KC, DeGue S, Niolon PH, Bishop J, Titus T, Noursi S, Dickerson SA, Whitaker D, Swider S, Remington P; Community Preventive Services Task Force. Intimate Partner and Sexual Violence Prevention Among Youth: A Community Guide Systematic Review. Am J Prev Med. 2022 Jan;62(1):e45-e55. doi: 10.1016/j.amepre.2021.06.021. Epub 2021 Nov 10. PMID 34772564
- [Background] Amar AF, Tuccinardi N, Heislein J, Simpson S. Friends Helping Friends: a nonrandomized control trial of a peer-based response to dating violence. Nurs Outlook. 2015 Jul-Aug;63(4):496-503. doi: 10.1016/j.outlook.2015.01.004. Epub 2015 Feb 3. PMID 26187089
- [Background] Jouriles EN, Krauss A, Vu NL, Banyard VL, McDonald R. Bystander programs addressing sexual violence on college campuses: A systematic review and meta-analysis of program outcomes and delivery methods. J Am Coll Health. 2018 Aug-Sep;66(6):457-466. doi: 10.1080/07448481.2018.1431906. Epub 2018 Mar 12. PMID 29405865
- [Background] Amar AF, Sutherland M, Kesler E. Evaluation of a bystander education program. Issues Ment Health Nurs. 2012 Dec;33(12):851-7. doi: 10.3109/01612840.2012.709915. PMID 23215986
- [Background] Barroso-Corroto E, Cobo-Cuenca AI, Laredo-Aguilera JA, Santacruz-Salas E, Pozuelo-Carrascosa DP, Rodriguez-Canamero S, Martin-Espinosa NM, Carmona-Torres JM. Dating violence, violence in social networks, anxiety and depression in nursing degree students: A cross-sectional study. J Adv Nurs. 2023 Apr;79(4):1451-1463. doi: 10.1111/jan.15170. Epub 2022 Feb 7. PMID 35128718
- See also: Word Health Organization. (2021). Violence against women — https://www.who.int/news-room/fact-sheets/detail/violence-against-women